CLINICAL TRIAL: NCT02879045
Title: The Effect of Elasticity Belly® Oil and Clarins® Tonic Body Treatment Oil in Prevention of Striae Gravidarum: A Randomized Controlled Clinical Trial
Brief Title: Comparison of 2 Body Oil in Prevention of Striae Gravidarum
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changning Maternity & Infant Health Hospital (Other)
Collaborators: Tongji University (Other)
Responsible Party: Principal Investigator, Ling Yang, associal professor, Shanghai Changning Maternity & Infant Health Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHCMIHH2016001
Record Dates: First submitted 2016-08-20; First posted 2016-08-25 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Prevention Harmful Effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- elasticity Belly® oil (Experimental): Volunteer's abdomen skin are divided two parts through medioventral line, half of the abdomen skin will apply the elasticity Belly® oil
  Interventions: Other: Elasticity Belly® oil

INTERVENTIONS:
Other: Elasticity Belly® oil — We will enroll about 50 Nulliparous women randomly, who are in their second trimester of pregnancy. We divide each of the volunteer's abdomen skin into two parts through medioventral line, one of the abdomen skin will receive the elasticity Belly® oil to prevent striae gravidarum, and the other side will use the Clarins® oil. Volunteers apply these two kinds of oil daily until birth. We'll take abdomen pictures before and after interventions, and the occurrence of striae on abdominal skin and its severity will be evaluated as our primary end point of the study.

SUMMARY:
The effect of elasticity Belly® oil and Clarins® Tonic Body Treatment Oil in prevention of striae gravidarum: A randomized controlled clinical trial.

DETAILED DESCRIPTION:
Objective: To compare the clinical efficacy of Elasticity Belly® oil and Clarins® Tonic Body Treatment Oil on the occurrence and severity of striae gravidarum.

Design: Parallel randomized controlled clinical trial. Setting: Gynaecology and Obstetrics department, Shanghai Changning Maternity and Infant Health Hospital, China Interventions: We will enroll about 50 Nulliparous women randomly, who are in their second trimester of pregnancy. Volunteer's abdomen skin are divided into two parts through medioventral line, half of the abdomen skin will receive the elasticity Belly® oil to prevent striae gravidarum, and the other side will use the Clarins® Tonic Body Treatment Oil. Volunteers apply these two kinds of oil daily until gestational age of 38-40 weeks. We'll take abdomen pictures before and after interventions, and the occurrence of striae on abdominal skin and its severity will be evaluated as our primary outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous females
* gestational age of 14-20 weeks
* 20 to 35 years old
* body mass index (BMI) from 18.5 to 25
* Clear consciousness, intelligence is normal,stable vital signs
* Voluntary participation, and sign the informed consent

Exclusion Criteria:

* allergy to skin care products
* twin pregnancies or polypregnancies
* polyhydramnios
* miscarriages
* development of a skin disease
* corticosteroid usage
* application of any other cream on the abdominal skin
* did not received allocated intervention
* drop out or lost to follow-up

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
occurrence and severity of striae gravidarum | second trimester to term birth
  volunteer's abdomen skin are divided into two parts through medioventral line, half of the abdomen skin will receive the elasticity Belly® oil , and the other side will use the Clarins® Tonic Body Treatment Oil. Volunteers apply these two kinds of oil daily until birth. We'll take abdomen pictures before and after interventions, and the occurrence of striae on abdominal skin and its severity will be evaluated as our primary end point of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shating Lei, PhD, Principal Investigator — Tongji University
Locations (1):
- Shanghai Changning Maternity & Infant Health Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No